CLINICAL TRIAL: NCT00258336
Title: Phase II Trial of Maintenance Rituximab Plus FavId® and GM-CSF Immunotherapy in Patients With Treatment-Naive Indolent B-Cell Lymphoma
Brief Title: Rituximab, Vaccine Therapy, and GM-CSF in Treating Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Favrille (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000449719; FAV-ID-70; FAV-ID-LYM-31
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2008-08

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; sargramostim

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine
Biological: rituximab
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Vaccines made from a person's cancer cells may help the body build an effective immune response to kill cancer cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving rituximab together with vaccine therapy and GM-CSF may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with vaccine therapy and GM-CSF works in treating patients with indolent B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of immunotherapy comprising rituximab, autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId™), and sargramostim (GM-CSF), in terms of response rate (partial and complete) and event-free survival, in patients with indolent B-cell non-Hodgkin's lymphoma.
* Determine the safety of this regimen in these patients.
* Evaluate development of an immune response in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

* Induction therapy: Patients receive rituximab IV over 2-4 hours once weekly for 4 weeks. Patients are evaluated for response at month 3. Patients with responding or stable disease proceed to maintenance therapy. Patients with progressive disease are removed from study.
* Maintenance therapy: Patients receive rituximab as in induction therapy in months 7, 13, and 19. Patients also receive autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId™) subcutaneously (SC) once on day 1 and sargramostim (GM-CSF) SC once daily on days 1-4 in months 4-6, 8-11, 14, 16, 18, 20, 22, and 24. Patients with continued response after completing 2 years of therapy may continue to receive FavId™ and GM-CSF once every 3 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed indolent B-cell non-Hodgkin's lymphoma of 1 of the following subtypes:

  * Grade 1 or 2 follicular lymphoma
* Tumor must be accessible to biopsy or biopsy material available for preparation of autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId™)
* Measurable or evaluable disease after node biopsy
* No mantle cell, marginal zone, MALT-type, small lymphocytic, or grade 3 follicular (follicular large cell) lymphoma
* No CNS involvement with lymphoma

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count > 100,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 2 times upper limit of normal
* Bilirubin ≤ 2 mg/dL

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* HIV negative
* No other medical or psychiatric disease that would preclude study compliance
* No other malignancy (active or treated) within the past 5 years

PRIOR CONCURRENT THERAPY:

Radiotherapy

* Prior local radiotherapy allowed

Other

* No other prior anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2004-08; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Event-free survival by Kaplan-Meier

SECONDARY OUTCOMES:
Overall response rate (partial and complete response) at month 6 and any time
Time-to-progression by Kaplan-Meier
Duration of response
Immune response by cellular or humoral anti-idiotype response positive
Safety

CONTACTS AND LOCATIONS:
Overall Officials: John F. Bender, PharmD, Study Chair — Favrille
Locations (1):
- Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee, United States